CLINICAL TRIAL: NCT00788606
Title: Feasibility Study of R-CHOP Plus Bevacizumab in Patients With Diffuse Large B Cell Lymphoma (DLBCL)
Brief Title: R-CHOP-B Bevacizumab for Diffuse Large B Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Toxicity and efficacy data from another trial
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR 2719
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Non-Hodgkin's Lymphoma; B-cell Lymphoma
Keywords: diffused large B cell lymphoma, DLBCL, R-Chop, bevacizumab; Diffuse large B-cell non-Hodgkin's lymphoma.
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — Bevacizumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab and Rituximab (Experimental): This study evaluates the feasibility using the anti-VEGF drug, bevacizumab, in combination with the standard treatment Rituximab in patients with stage II, III and IV diffuse large B cell lymphoma (DLBCL)
  Interventions: Drug: bevacizumab, Rituximab

INTERVENTIONS:
Drug: bevacizumab, Rituximab — 6 cycles of treatment. Bevacizumab at a dose of 15 mg/kg, diluted in normal saline will be administered as a intravenous infusion over 30 to 90 minutes on Day 1 of each cycle. Rituzimab 375 mg/m2 is given as a intravenous infusion after the administration of prednisolone and before the other cytotoxic drugs on Day 1 of each cycle.

SUMMARY:
This study evaluates the use of the standard treatment R-CHOP plus the anti-VEGF drug, bevacizumab and whether this treatment is feasible in patients with stage II, III and IV diffuse large B cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
Non-Hodgkin's lymphoma is increasing in incidence with more than 287,000 cases world-wide and 9000 cases in UK diagnosed each year. DLBCL is the most frequently occurring NHL, constituting approximately 31% of all non-Hodgkin's lymphomas.

Rituximab-CHOP chemotherapy has shown clinical efficacy and is regarded as standard treatment in patients with DLBCL. NICE has recently approved the use of rituzimab in combination with CHOP for all newly diagnosed patients with DLBCL stage II-IV.

Angiogenesis plays an important role in the pathophysiology of both solid tumours and hematologic malignancies. Vascular endothelial growth factor (VEGF) is the most important pro-angiogenic factor involved in normal and pathologic angiogenesis and studies have also implicated VEGF in lymphomagenesis. Elevated VEGF gene expression correlates with diffuse large B cell lymphoma subtypes of poor prognosis on microarray analysis. In patients with lymphoma, high circulating serum VEGF levels have been strongly associated with poor clinical outcomes independent of other predictive factors.

Bevacizumab is a humanized monoclonal antibody that binds to VEGF thus preventing binding to its receptors thus inhibiting the downstream pathways dependent on receptor stimulation. Bevacizamab has shown activity in solid tumours (colorectal, renal, breast and non-small cell lung cancer) and early results suggest that the combination of R-CHOP plus bevacizamab is feasible in patients with non Hodgkin's lymphoma.

Patients will be treated with a minimum of 6 cycles of treatment. A further 2 cycles, to a total of 8 cycles, may be administered if continuing response to treatment has been documented but residual disease is still detectable on restaging after 6 cycles. Each cycle of treatment is 21 days.

Follow up - a) Clinic visit with physical examination at 3, 6, 9, 12, 18 and 24 months after completion of R-CHOP-B, then annually.

b) CT scan of chest, abdomen and pelvis at 3 months and 1 year after finishing treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Histological proven diffuse large B cell non-Hodgkin's lymphoma (DLBCL) according to the World Health Organization classification including morphological variants. The B cell nature of the proliferation must be verified by the positivity with an anti-CD20 antibody. All histology will be reveiwed by a central Lymphoma Trials Office pathology panel.
* No previous chemotherapy, radiotherapy or other investigational drug for this indication.
* Stage II, III and IV disease.
* WHO performance status 0<2.
* Adequate bone marrow function with platelets > 100x109/l: neutrophils > 1.5x109/l at the time of study entry unless attributed to bone marrow infiltration by lymphoma.
* Serum creatinine < 150μmol/l , serum bilirubin < 35μmol/l and transaminases < 2.5 x upper limit of institutional normal range unless attributed to lymphoma.
* Normal MUGA or echocardiogram without any areas of abnormal contractility. Patients must have an acceptable left ventricular ejection fraction (LVEF) > 50%.
* No current uncontrolled medical condition.
* No active malignant disease other than basal or squamous cell carcinoma of the skin or carcinoma in situ of the uterine cervix in the last 10 years.
* Adequate contraceptive precautions for all patients of childbearing potential.
* Written, informed consent.

Exclusion Criteria:

* T-cell lymphoma or transformed follicular lymphoma.
* Previous history of treated or non-treated indolent lymphoma. However, patients not previously diagnosed who have a large B-cell lymphoma with some small cell infiltration in bone marrow or lymph node may be included.
* Past history of heart failure or uncontrolled angina pectoris.
* Central nervous system, meningeal involvement or cord compresssion by the lymphoma
* Cardiac contra-indication to doxorubicin (abnormal contractility on echocardiography or nuclear medicine examination[MUGA])
* Neurological contra-indication to vincristine (e.g pre-existing diabetic neuropathy).
* Any other serious active disease
* General status that does not allow the administration of 8 courses of CHOP according to the investigator
* Positive serology for HIV, Hepatitis B or Hepatitis C
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent
* Bevacuzumab related criteria:

  * No major surgery, major trauma or open biopsy within 28 days prior to study entry. Patients requiring insertion of central venous access for treatment (e.g due to poor venous access) should have the procedure performed at least 2 days before starting treatment.
  * No serious, non-healing would, ulcer or bone fracture.
  * Absence of obvious risk of requiring emergency surgery after commencement of study treatmene, such as impending bowel obstruction.
  * Absense of clinically significant (i.e active) cardiovascular disease e.g. cerebrovascular accidents (<6 months prior to randomisation), myocardial infarction (< 1 year prior to randomisation), uncontrolled hypertension while receiving chronic medication, unstable angina, New York Hearth Association (NYHA) grade II or greater congestive heart failure, or serious cardiac arrhymia requiring medication.
  * No recent history of any active gastrointestinal inflammatory condition such a peptic ulcer disease, diverticulitis or inflammatory bowel disease. If patients have a known diagnosis of any of the above, evidence of disease control is required by negative endoscopy within the last 28 days.
  * No evidence of bleeding disthesis or coagulopathy.
  * No recent commencement of full oral anticoagulation (warfarin), unless stable and within therapeutic range for at least 10 days. No thrombolytic therapy within 10 days prior to commencement of study treatment.
  * No chronic, daily treatment with high-dose aspirin (> 325mg/day) or nonsteroidal anti-inflammatory medications (those known to inhibit platelet function at doses used to treat chronic inflammatory diseases).
  * No chronic treatment with corticosteriods (dose of . 10 mg/day methylprednisolone equivalent) (excluding inhaled steroids).
  * No known allergy to Chinese hamster ovary cell proteins or other recombinant human or humanized antibodies or to any other excipients of bevacizumab formulation, platinum compounds or to any other components of the study drugs.
  * No proteinuria at baseline as defined by>1g of protein/24 hr by 24-hour urine collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is cardiac and bevacizumab-specific toxicity. Toxicities will be evaluated according to the NCI Common Toxicity Criteria for Adverse Events v3.0 | 1 year

SECONDARY OUTCOMES:
Response rates, failure free survival, and overall survival will be evaluated and are secondary endpoints | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - David Cunningham, Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Royal Marsden NHS Foundation Trust, Sutton, Surrey